CLINICAL TRIAL: NCT06688136
Title: Ultrasound-guided Transmuscular Quadratus Lumborum and Modified Erector Spinae Plane Block Versus Periarticular Infiltration for Pain Management After Total Hip Arthroplasty
Brief Title: QLESP Block Versus Periarticular Infiltration for Postoperative Analgesia in Hip Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xi Wu, Huazhong University of Science and Technology, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: WHUH20241101
Record Dates: First submitted 2024-11-11; First posted 2024-11-14 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2024-11

CONDITIONS: Regional Anaesthesia
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- transmuscular quadratus lumborum and modified erector spinae plane (QLESP) block (Experimental): Twenty ml of 0.4% ropivacaine was administered between the erector spinae muscle and the transverse process. Twenty ml of 0.4% ropivacaine was subsequently given between the quadratus lumborum and the psoas major muscles.
  Interventions: Drug: ropivacaine
- Infiltration (Active Comparator): Periarticular infiltration of 40 ml of 0.4% ropivacaine prior to closing the incision
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: ropivacaine — Ropivacaine 200 mg diluted to 50 mL

SUMMARY:
Local and/or regional analgesia techniques are critical components of an optimal multimodal analgesia technique, as they have been shown to improve pain relief as well as reduce opioid requirements. Optimal pain management technique balances pain relief with concerns about safety and adverse effects associated with analgesic techniques. Periarticular infiltration (PAI) is increasingly included as a component of multimodal analgesia technique for patients undergoing THA, as it provides improved postoperative pain relief with no effects on quadriceps function. Recently, our group has developed a novel transmuscular quadratus lumborum and modified erector spinae plane (QLESP) block, which is characterized by simple operation, high efficiency, and wide dermatomal coverage of sensory block. Therefore, we designed a randomized controlled trial to compare ultrasound-guided QLESP with PAI as a component of non-opioid analgesic regimen in patients undergoing THA via posterior approach. We hypothesized that QLESP would provide superior analgesia when compared with PAI. The primary outcome of the study was postoperative opioid requirements within the initial 24-h postoperative period after THA. The secondary objectives were to compare pain scores, postoperative quadriceps strength, the time to first rescue analgesia, opioid-related adverse effects, time to ambulation, and the time to hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 yrs
2. American Society of Anesthesiologists classification 1-3
3. Body mass index between 20 and 35 (kg/m2)
4. Undergo elective primary unilateral THA via a posterolateral approach
5. Informed consent

Exclusion Criteria:

1. A known allergy to the drugs being used
2. Pre-existing neuropsychiatric disorders or language barrier
3. Analgesics intake, history of substance abuse
4. Contraindications to peripheral nerve block
5. Acute cerebrovascular disease
6. Severe liver failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
The cumulative opioid consumption | At 24 postoperative hours

SECONDARY OUTCOMES:
The pain scores determined by the numeric rating scale (NRS, 0-10) | Postoperative 48 hours
Quadriceps strength | Postoperative 48 hours
Postoperative hospital length of stay | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xi Wu, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No